CLINICAL TRIAL: NCT04574245
Title: Retrospective Multi-institutional Cohort Study of Gastric Cancer Liver Metastasis in Real-world Data of China
Brief Title: Gastric Cancer Liver Metastasis Cohort of China
Acronym: RECORD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Lin Chen, Prof., Chinese PLA General Hospital
Other Study IDs: S2020-381
Record Dates: First submitted 2020-09-23; First posted 2020-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Stomach Neoplasms; Neoplasm Metastasis
Keywords: Prognosis; Multidisciplinary treatment; C-GCLM Classification; Gastric cancer; Liver metastasis
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — Gastrectomy; Hepatectomy; Radiofrequency Ablation; Drug Therapy; Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Resectable group
  Interventions: Procedure: Gastrectomy; Hepatectomy
- Potentially resectable group
- Unresectable group

INTERVENTIONS:
Procedure: Gastrectomy; Hepatectomy
  Other Names: Radiofrequency ablation; Chemotherapy; Immunotherapy; Target therapy
  Groups: Resectable group

SUMMARY:
This multi-institutional retrospective cohort study aimed to describe and analyze the overall clinical characteristics, therapeutic status and prognosis pattern of gastric cancer liver metastasis (GCLM) in China.

ELIGIBILITY:
Inclusion Criteria:

* Gastric cancer liver metastases cases aged over 18 years old;
* Primary gastric carcinoma (including different histopathological types) confirmed by biopsy or surgery (pre-, intra- or post- treatment);
* In hospital cases between 2020/01/01 to 2019/12/3.

Exclusion Criteria:

* Poor compliance to treatment or lost to follow-up;
* Gross loss of clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible in-hospital gastric cancer liver metastases cases.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year overall survival | 2011/01/01-2020/12/31
  The proportion (%) of gastric cancer liver metastasis patients that survived beyond one-year follow-up period.
3-year overall survival | 2011/01/01-2021/12/31
  The proportion (%) of gastric cancer liver metastasis patients that survived beyond three-year follow-up period.
5-year overall survival | 2011/01/01-2021/12/31
  The proportion (%) of gastric cancer liver metastasis patients that survived beyond five-year follow-up period.

SECONDARY OUTCOMES:
The incidence of gastric cancer liver metastasis cases | 2010/01/01-2019/12/31
  The rate of gastric cancer liver metastasis cases divided by all gastric cancer cases in the study period.
The proportion for synchronous and metachronous liver metastases cases | 2010/01/01-2019/12/31
  The proportion (%) of synchronous or metachronous gastric cancer liver metastases cases in all gastric cancer cases
The survival of patients that recieved different therapeutic methods | 2010/01/01-2019/12/31
  The proportion (%) of patients under different therapies that survived beyond specific follow-up period.
The prognostic predictive value for patients with different C-GCLM classification | 2010/01/01-2019/12/31
  The proportion (%) of patients of different classification that survived beyond specific follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- General Surgery Institute, China PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang K, Chen L. Chinese consensus on the diagnosis and treatment of gastric cancer with liver metastases. Ther Adv Med Oncol. 2020 Feb 20;12:1758835920904803. doi: 10.1177/1758835920904803. eCollection 2020. PMID 32127925